CLINICAL TRIAL: NCT06749431
Title: MERCuRE (MEniscus, Restoration, Conservation, and Repair) Group Study on Clinical Outcomes, Graft Longevity, and Chondral Protection Following Primary or Revision Meniscal Allograft Transplantation Surgery
Brief Title: Clinical Outcomes, Graft Longevity, and Chondral Protection Following Primary or Revision Meniscal Allograft Transplantation Surgery
Status: Enrolling by invitation | Type: Observational
Sponsor: Joint Restoration Foundation, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 001
Record Dates: First submitted 2024-11-08; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Meniscus Tear; Meniscus Disorder; Patient Satisfaction
Keywords: Meniscal Allograft Transplant
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years

SUMMARY:
The MERCuRE (MEniscus, REstoration, Conservation, and Repair) group is embarking on a 20-year follow-up study to evaluate the clinical outcomes, graft longevity, and chondral protection following primary or revision Meniscal Allograft Transplantation surgery This clinical investigation is a prospective, primary observational, open-label, non-randomized, multi-center study. It is designed to collect clinical follow-up data on patients

ELIGIBILITY:
Inclusion Criteria:

Subjects enrolled in this study must meet all of the following inclusion criteria:

* Males and females aged 10-65 years
* MRI or arthroscopic images confirming the suitability for meniscus transplantation.
* Patients undergoing an isolated primary/revision MAT (meniscal allograft transplant) procedure, or concomitant MAT with other knee procedures such as ligament reconstruction, realignment osteotomy, or cartilage resurfacing.
* Medically suitable for meniscus transplantation.
* Appropriate understanding of the language of the surgical center in terms of communication and reading.
* Ability of the Patient or parent/guardian to provide informed consent.

Exclusion Criteria:

* Inability to comply with rehabilitation programs.
* Patient aged less than 10 years and more than 65.
* Presence of diffuse full thickness cartilage loss (widespread ICRS Grade III-IV chondral damage) and/or architectural remodeling of bone (i.e. flattening of condyle) in the knee of interest.
* Significant medical comorbidities that limit patients from undergoing surgery.
* Presence of confounding neuromuscular, genetic/congenital, or post-traumatic conditions.

Ages: 10 Years to 65 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with meniscal deficiency
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-01-05 (Estimated); Primary Completion 2030-01-05 (Estimated); Study Completion 2050-01-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of PROM: The Knee Injury and Osteoarthritis Outcome (KOOS) Score | 3 months, 6 months, 1 year, 2 years, 5 years, 10 years, 15 years, and 20 years post-operatively
  Evaluation of knee symptoms and function, reported on a scales from 0 to 100 where 0 represents extreme knee problems and 100 represents no knee problems.
Evaluation of PROM: Marx activity rating scale for patients > 18 years old | 3 months, 6 months, 1 year, 2 years, 5 years, 10 years, 15 years, and 20 years post-operatively
  Measure of activities associated with high level knee function within the last year, scored from 0 to 16 where 0 is activities less than one time in a month and 16 is activities 4 or more times in a week.
Evaluation of PROM: Pediatric Functional Activity Brief Scale (Pedi-FABS) score for patients 10-18 years old | 3 months, 6 months, 1 year, 2 years, 5 years, 10 years, 15 years, and 20 years post-operatively
  Measure of activity within the last month, scored from 0-30 where 0 is participating in activities less than one time per month and 16 is participating in activities more than 4 times per week.
Evaluation of PROM: Western Ontario Meniscal Evaluation Tool (WOMET) score | 3 months, 6 months, 1 year, 2 years, 5 years, 10 years, 15 years, and 20 years post-operatively
  Measure of health-related quality of life for meniscus symptoms, scored from 0 to 100 where 0 is no physical symptoms or emotional feeling and 100 is extreme symptoms and extreme emotional feeling.
Clinical Success | Through study completion, up to 20 years post-operatively.
  Data on failure defined as removal of the whole or large portion of the graft (total or subtotal meniscectomy or a large irreparable radial tear), conversion to arthroplasty or revision of the meniscal transplant.
Serial Imaging: Radiographs | baseline (pre-op), 3 months, 6 months, 1 year, 2 years, 5 years, 10 years, 15 years, and 20 years post-operatively
  Knee radiographs to determine graft longevity, status/presence of extrusion and the post-operative chondral status of the knee.
Serial Imaging: Ultrasound | baseline (pre-op), 3 months, 6 months, 1 year, 2 years, 5 years, 10 years, 15 years, and 20 years post-operatively
  Knee ultrasound to determine graft longevity, status/presence of extrusion and the post-operative chondral status of the knee.
Serial Imaging: Magnetic Resonance Imaging (MRI) | baseline (pre-op), 3 months, 6 months, 1 year, 2 years, 5 years, 10 years, 15 years, and 20 years post-operatively
  Knee MRI to determine graft longevity, status/presence of extrusion and the post-operative chondral status of the knee.

SECONDARY OUTCOMES:
Minimal Clinically Important Difference (MCID) in Patient Reported Outcomes (PROs) | Calculated by anchor question response pre-operatively, 6 months, 1 year, 2 years, 5 years, 10 years, 15 years, and 20 years post-operatively.
  To define the Minimal Clinically Important Difference (MCID) for the above mentioned PRO's in these patients, and to correlate patients' demographics and surgical status of the knee, to the MCID.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Health, Plano, Texas, United States